CLINICAL TRIAL: NCT06739746
Title: Research on the Sources of Noise in Post Anesthesia Care Unit and the Impact of Noise on Medical Staff
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Shenzhen Mindray Bio-Medical Electronics Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Min Su, Director, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2024-214-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-12

CONDITIONS: Noise Exposure
Keywords: Noise; Post anesthesia care unit; Medical staff

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Medical staff group: Investigate the demographic information and subjective perception of noise among medical staff in the post anesthesia care unit.
  Interventions: Other: No intervention measures
- Hospital Group: Investigate the staffing, size, number of beds, noise levels, etc. of post anesthesia care unit in different hospitals.
  Interventions: Other: No intervention measures

INTERVENTIONS:
Other: No intervention measures — No intervention measures

SUMMARY:
The study aims to clarify the sources and influencing factors of noise in the post anesthesia care unit, as well as the perception of noise by medical staff through survey table, in order to improve the noise environment, optimize noise management, protect medical staff, and enhance medical quality.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as nurses, doctors, or technicians in the Post Anesthesia Care Unit;
* Have at least continuous 6 months of work experience in the Post Anesthesia Care Unit;
* Able to read and answer questionnaires in Chinese fluently.

Exclusion Criteria:

* Have hearing impairments or other conditions affecting auditory perception;
* Have participated in similar studies and completed related surveys within the past 6 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical staff in the post anesthesia care unit
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Main noise decibel | From enrollment to the end of observation at 1 week
  The level of noise decibel in the post anesthesia care unit when the number of patients is between half and three-quarters of the total number of beds. Using noise vibration measuring instrument (AWA5688, Hangzhou Aihua Instrument Co., Ltd.) to measure the noise decibel.

SECONDARY OUTCOMES:
Secondary noise decibel | From enrollment to the end of observation at 1 week
  The level of noise decibel in the post anesthesia care unit when the number of patients is not between half and three-quarters of the total number of beds. Using noise vibration measuring instrument (AWA5688, Hangzhou Aihua Instrument Co., Ltd.) to measure the noise decibel.
Area of post anesthesia care unit | From enrollment to the end of observation at 1 week
  Measure the area of the post anesthesia care unit using a tape measure, in square meters.
Number of beds of post anesthesia care unit | From enrollment to the end of observation at 1 week
Medical personnel allocation situation | From enrollment to the end of observation at 1 week
  Number of anesthesiologists and nurses
Staying time in post anesthesia care unit of patients | From enrollment to the end of observation at 1 week
Number of patients with or without tracheal intubation retained | From enrollment to the end of observation at 1 week
  Defined as patients whether retaining the endotracheal tube before entering the post anesthesia care unit
Daily working hours of medical staff | From enrollment to the end of observation at 1 week
Working years of medical staff | From enrollment to the end of observation at 1 week
Subjective perception of noise by medical personnel | From enrollment to the end of observation at 1 week
  Using multiple-activity scale for hyperacusis (MASH) that is proposed by Dauman in 2005 to evaluate emotion. MASH categorizes the level of annoyance caused by noise into five levels: absent, mild, moderate, substantial, and severe. In our study, every individuals will be given a score of zero to four based on this five levels, higher scores mean a worse outcome.
The impact of noise on the work of medical personnel | From enrollment to the end of observation at 1 week
  Based on our preliminary research findings, we have made a questionnaire titled "Working Conditions in Noisy Environments", which indicates that the impact of noise in the post anesthesia care unit on the work of medical personnel is usually as follows: no impact, failure to hear patient calls or needs in a timely manner, inability to identify alarms from specific medical equipment, need to speak loudly, and throat discomfort.
The source of noise as perceived by the medical staff | From enrollment to the end of observation at 1 week
  Based on our preliminary research findings, we have made a questionnaire titled "Noise source in Post Anesthesia Care Unit", which includes monitor, sputum suction device, ventilator, conversation, mobile phone, printer, outdoor factors (such as the move of transfer beds.), and other.
Satisfaction of medical staff with the current noise situation | From enrollment to the end of observation at 1 week
  Based on our preliminary research findings, we have made a questionnaire titled "Satisfaction with the Current Noise Situation in the Post Anesthesia Care Unit", which includes very satisfied, satisfied, general,dissatisfied, and very dissatisfied.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR